CLINICAL TRIAL: NCT05780788
Title: Characterizing Orthodontic Tooth Movement in Real Time Using Dental Monitoring Scans: a Pilot Study
Brief Title: Characterizing Orthodontic Tooth Movement With Photographic Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Flavio Uribe, Associate Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-113-2
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Canine Retraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Canine retraction arm (Experimental): Canine retraction
  Interventions: Device: Monitoring Tooth Movement

INTERVENTIONS:
Device: Monitoring Tooth Movement — Monitoring Canine Retraction

SUMMARY:
Characterizing orthodontic tooth movements in real time by using photographic scans to monitor teeth movement. The photographic scans will also be compared to 3D model scans. Canine retraction over the course of 1 orthodontic visit will be measured.

DETAILED DESCRIPTION:
The accuracy and reliability of Dental Monitoring scans is be evaluated and compared to that of iTero digital scans during maxillary canine retraction. The magnitude and type of tooth movement occurring in a one month period in patients undergoing maxillary canine retraction will be measured. Patients undergoing orthodontic treatment in the Center for Orthodontic Care at UConn Health will be evaluated for the inclusion criteria. A total of twenty patients whose orthodontic treatment plan required extraction of at least one premolar in the maxillary arch will be recruited. The patient will be required to take photographs and video scans as dictated by Dental Monitoring (DM) on the first and final days of the study period (four weeks), while iTero scans are taken by the provider in clinic on these same days. Patient will also be periodically taking photographic scans at home using Dental Monitoring. The DM scans taken by the patient will be compared to the iTero digital scans taken by the provider. This can be done by superimposing the stereolithographic (STL) files created from each scan and assessing the amount of deviation between the 3D models. The types of tooth movement occurring during canine retraction in buccolingual, mesiodistal, and incisogingival planes will be quantified using Doctor Dashboard software available in DM. DM's 3D matching technology allows superimposition of teeth from each 3D model created per scan. Each tooth and its movements are graphed in a detailed manner to provide precise information about its type of movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fixed orthodontic appliances
* Treatment plan requiring extraction of at least one maxillary premolar
* Male and female
* Permanent dentition from first molar to first molar in the maxilla
* Teeth with normal crown morphology
* Fully erupted canines
* Above 11 years of age
* Patients with any cellular phone with a camera

Exclusion Criteria:

* Lack of extraction in orthodontic treatment plan
* Syndromic patients
* Cleft lip/palate patients
* Removable appliances

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Uribe, DDS, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects that were consented participated in the study
Period: Overall Study
Arm/Group | Canine retraction arm
Started | 36
Completed | 22
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: A total of 36 participants were enrolled, but only 22 had usable baseline data.
Arm/Group | Canine Retraction Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants] — Population: The number of patients analyzed was based on usable data. Specifically, scans that were not of appropriate quality for measurements were excluded.
  Participants
    <=18 years | 17
    Between 18 and 65 years | 5
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of patients analyzed was based on usable data. Specifically, scans that were not of appropriate quality for measurements were excluded.
  years | 17.41 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number of patients analyzed was based on usable data. Specifically, scans that were not of appropriate quality for measurements were excluded.
  Participants
    Female | 16
    Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The number of patients analyzed was based on usable data. Specifically, scans that were not of appropriate quality for measurements were excluded.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 6
    White | 6
    More than one race | 0
    Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants] — Population: The number of patients analyzed was based on usable data. Specifically, scans that were not of appropriate quality for measurements were excluded.
  Participants
    United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Between Patient-taken DM Scan and Provider-taken iTero Scan
Description: Deviation between the photographic and intraoral scan will be measured via root mean square (RMS) in millimeters (mm).
Time Frame: Initial Deviation T0 (Baseline), Final Deviation T9 (34-37 days)
Population: A total of 36 participants were enrolled in the study. Due to scan quality issues, only 22 participants had usable data for analysis. Specifically, 13 participants were analyzed for the Initial Deviation outcome, and 15 participants for the Final Deviation outcome.
Measure: Median (Inter-Quartile Range); unit: Millimeters (mm)
Arm/Group | Canine retraction arm
Number analyzed (Participants) | 22
Millimeters (mm)
  Initial Deviation T0 (Baseline): number analyzed (Participants) | 13
  Initial Deviation T0 (Baseline) | 0.0001 [0.0001 to 0.0005]
  Final Deviation T9 (34-37 days): number analyzed (Participants) | 15
  Final Deviation T9 (34-37 days) | 0.0500 [0.0400 to 0.0600]

2. Secondary Outcome: Tracking Maxillary Canine Tooth Movement (Displacement)
Description: Magnitude of canine tooth movement for every 4-5 days during a one month period. Measurements will be done in mm in three planes of space. Measurement reported in mm at each timepoint is the cumulative movement up to that timpoint during the one month of monitoring of tooth movement.
Time Frame: T1 (3-5 days), T2 (6-9 days), T3 (10-13 days), T4 (14-17 days), T5 (18-21 days), T6 (22-25 days), T7 (26-29 days), T8 (30-33 days), T9 (34-37days).
Population: A total of 36 participants were enrolled, but only 21 had usable data due to scan quality issues. Each tooth (canine and molar on both sides) was analyzed individually, and analysis could vary by side. Sample sizes varied by tooth and time point depending on image availability.
Measure: Median (Inter-Quartile Range); unit: Millimeters
Arm/Group | Canine retraction arm
Number analyzed (Participants) | 21
Millimeters
  Right canine displacement movement in x- axis (anteroposterior)T1 (3-5 days): number analyzed (Participants) | 17
  Right canine displacement movement in x- axis (anteroposterior)T1 (3-5 days) | -0.36 [-0.46 to -0.15]
  Right canine displacement movement in y- axis (vertical) T1 (3-5 days): number analyzed (Participants) | 17
  Right canine displacement movement in y- axis (vertical) T1 (3-5 days) | -0.06 [-0.09 to -0.03]
  Right canine displacement movement in z- axis (transverse) T1 (3-5 days): number analyzed (Participants) | 17
  Right canine displacement movement in z- axis (transverse) T1 (3-5 days) | -0.03 [-0.14 to 0.01]
  Left canine displacement movement in x- axis (anteroposterior) T1 (3-5 days): number analyzed (Participants) | 17
  Left canine displacement movement in x- axis (anteroposterior) T1 (3-5 days) | -0.39 [-0.54 to -0.26]
  Left canine displacement movement in y- axis (vertical) T1 (3-5 days): number analyzed (Participants) | 17
  Left canine displacement movement in y- axis (vertical) T1 (3-5 days) | -0.10 [-0.15 to -0.03]
  Left canine displacement movement in z- axis (transverse) T1 (3-5 days): number analyzed (Participants) | 17
  Left canine displacement movement in z- axis (transverse) T1 (3-5 days) | -0.13 [-0.23 to 0.01]
  Right canine displacement movement in x- axis (anteroposterior)T2 (6-9 days): number analyzed (Participants) | 16
  Right canine displacement movement in x- axis (anteroposterior)T2 (6-9 days) | -0.515 [-0.67 to -0.395]
  Right canine displacement movement in y- axis (vertical) T2 (6-9 days): number analyzed (Participants) | 16
  Right canine displacement movement in y- axis (vertical) T2 (6-9 days) | -0.07 [-0.12 to -0.05]
  Right canine displacement movement in z- axis (transverse) T2 (6-9 days): number analyzed (Participants) | 16
  Right canine displacement movement in z- axis (transverse) T2 (6-9 days) | -0.11 [-0.15 to -0.04]
  Left canine displacement movement in x- axis (anteroposterior) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine displacement movement in x- axis (anteroposterior) T2 (6-9 days) | -0.66 [-0.79 to -0.45]
  Left canine displacement movement in y- axis (vertical) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine displacement movement in y- axis (vertical) T2 (6-9 days) | -0.11 [-0.17 to 0.01]
  Left canine displacement movement in z- axis (transverse) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine displacement movement in z- axis (transverse) T2 (6-9 days) | -0.21 [-0.35 to -0.06]
  Right canine displacement movement in x- axis (anteroposterior)T3 (10-13days): number analyzed (Participants) | 15
  Right canine displacement movement in x- axis (anteroposterior)T3 (10-13days) | -0.52 [-0.80 to -0.28]
  Right canine displacement movement in y- axis (vertical) T3 (10-13 days): number analyzed (Participants) | 15
  Right canine displacement movement in y- axis (vertical) T3 (10-13 days) | -0.13 [-0.15 to -0.07]
  Right canine displacement movement in z- axis (transverse) T3(10-13 days): number analyzed (Participants) | 15
  Right canine displacement movement in z- axis (transverse) T3(10-13 days) | -0.07 [-0.11 to -0.02]
  Left canine displacement movement in x- axis (anteroposterior) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine displacement movement in x- axis (anteroposterior) T3 (10-13 days) | -0.82 [-0.97 to -0.57]
  Left canine displacement movement in y- axis (vertical) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine displacement movement in y- axis (vertical) T3 (10-13 days) | -0.14 [-0.21 to -0.01]
  Left canine displacement movement in z- axis (transverse) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine displacement movement in z- axis (transverse) T3 (10-13 days) | -0.21 [-0.39 to -0.05]
  Right canine displacement movement in x- axis (anteroposterior)T4 (14-17 days): number analyzed (Participants) | 16
  Right canine displacement movement in x- axis (anteroposterior)T4 (14-17 days) | -0.74 [-0.88 to -0.52]
  Right canine displacement movement in y- axis (vertical) T4 (14-17 days): number analyzed (Participants) | 16
  Right canine displacement movement in y- axis (vertical) T4 (14-17 days) | -0.14 [-0.21 to -0.07]
  Right canine displacement movement in z- axis (transverse) T4 (14-17 days): number analyzed (Participants) | 16
  Right canine displacement movement in z- axis (transverse) T4 (14-17 days) | -0.12 [-0.34 to -0.03]
  Left canine displacement movement in x- axis (anteroposterior) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine displacement movement in x- axis (anteroposterior) T4 (14-17 days) | -0.76 [-1.04 to -0.63]
  Left canine displacement movement in y- axis (vertical) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine displacement movement in y- axis (vertical) T4 (14-17 days) | -0.18 [-0.27 to -0.07]
  Left canine displacement movement in z- axis (transverse) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine displacement movement in z- axis (transverse) T4 (14-17 days) | -0.28 [-039 to -0.09]
  Right canine displacement movement in x- axis (anteroposterior)T5 (18-21 days): number analyzed (Participants) | 15
  Right canine displacement movement in x- axis (anteroposterior)T5 (18-21 days) | -0.82 [-1.04 to -0.58]
  Right canine displacement movement in y- axis (vertical) T5 (18-21 days): number analyzed (Participants) | 15
  Right canine displacement movement in y- axis (vertical) T5 (18-21 days) | -0.18 [-0.26 to -0.11]
  Right canine displacement movement in z- axis (transverse) T5 (18-21 days): number analyzed (Participants) | 15
  Right canine displacement movement in z- axis (transverse) T5 (18-21 days) | -0.16 [-0.40 to -0.03]
  Left canine displacement movement in x- axis (anteroposterior) T5 (18-21 days): number analyzed (Participants) | 15
  Left canine displacement movement in x- axis (anteroposterior) T5 (18-21 days) | -0.94 [-1.18 to -0.74]
  Left canine displacement movement in y- axis (vertical) T5 (18-21 days): number analyzed (Participants) | 15
  Left canine displacement movement in y- axis (vertical) T5 (18-21 days) | -0.17 [-0.33 to -0.05]
  Left canine displacement movement in z- axis (transverse) T5 (18 -21days): number analyzed (Participants) | 15
  Left canine displacement movement in z- axis (transverse) T5 (18 -21days) | -0.27 [-0.52 to -0.06]
  Right canine displacement movement in x- axis (anteroposterior)T6 (22-25 days): number analyzed (Participants) | 13
  Right canine displacement movement in x- axis (anteroposterior)T6 (22-25 days) | -0.98 [-1.17 to -0.72]
  Right canine displacement movement in y- axis (vertical) T6 (22-25 days): number analyzed (Participants) | 13
  Right canine displacement movement in y- axis (vertical) T6 (22-25 days) | -0.22 [-0.28 to -0.11]
  Right canine displacement movement in z- axis (transverse) T6 (22 -25days): number analyzed (Participants) | 13
  Right canine displacement movement in z- axis (transverse) T6 (22 -25days) | -0.21 [-0.55 to 0]
  Left canine displacement movement in x- axis (anteroposterior) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine displacement movement in x- axis (anteroposterior) T6 (22-25 days) | -1.14 [-1.28 to -0.86]
  Left canine displacement movement in y- axis (vertical) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine displacement movement in y- axis (vertical) T6 (22-25 days) | -0.22 [-0.37 to -0.10]
  Left canine displacement movement in z- axis (transverse) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine displacement movement in z- axis (transverse) T6 (22-25 days) | -0.30 [-0.60 to -0.06]
  Right canine displacement movement in x- axis (anteroposterior) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine displacement movement in x- axis (anteroposterior) T7 (26-29 days) | -0.99 [-1.29 to -0.68]
  Right canine displacement movement in y- axis (vertical) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine displacement movement in y- axis (vertical) T7 (26-29 days) | -0.23 [-0.36 to -0.16]
  Right canine displacement movement in z- axis (transverse) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine displacement movement in z- axis (transverse) T7 (26-29 days) | -0.24 [-0.46 to -0.03]
  Left canine displacement movement in x- axis (anteroposterior) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine displacement movement in x- axis (anteroposterior) T7 (26-29 days) | -1.16 [-1.36 to -0.93]
  Left canine displacement movement in y- axis (vertical) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine displacement movement in y- axis (vertical) T7 (26-29 days) | -0.22 [-0.35 to -0.19]
  Left canine displacement movement in z- axis (transverse) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine displacement movement in z- axis (transverse) T7 (26-29 days) | -0.30 [-0.57 to -0.06]
  Right canine displacement movement in x- axis (anteroposterior) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine displacement movement in x- axis (anteroposterior) T8 (30-33 days) | -1.08 [-1.43 to -0.66]
  Right canine displacement movement in y- axis (vertical) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine displacement movement in y- axis (vertical) T8 (30-33 days) | -0.32 [-0.40 to -0.18]
  Right canine displacement movement in z- axis (transverse) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine displacement movement in z- axis (transverse) T8 (30-33 days) | -0.30 [-0.58 to -0.06]
  Left canine displacement movement in x- axis (anteroposterior) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine displacement movement in x- axis (anteroposterior) T8 (30-33 days) | -1.29 [-1.67 to -1.01]
  Left canine displacement movement in y- axis (vertical) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine displacement movement in y- axis (vertical) T8 (30-33 days) | -0.32 [-0.53 to -0.24]
  Left canine displacement movement in z- axis (transverse) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine displacement movement in z- axis (transverse) T8 (30-33 days) | -0.42 [-0.75 to -0.30]
  Right canine displacement movement in x- axis (anteroposterior) T9 (34 -37days): number analyzed (Participants) | 7
  Right canine displacement movement in x- axis (anteroposterior) T9 (34 -37days) | -1.19 [-1.44 to -0.82]
  Right canine displacement movement in y- axis (vertical) T9 (34 -37days): number analyzed (Participants) | 7
  Right canine displacement movement in y- axis (vertical) T9 (34 -37days) | -0.35 [-0.56 to -0.18]
  Right canine displacement movement in z- axis (transverse) T9 (34 -37days): number analyzed (Participants) | 7
  Right canine displacement movement in z- axis (transverse) T9 (34 -37days) | -0.24 [-0.75 to -0.08]
  Left canine displacement movement in x- axis (anteroposterior) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine displacement movement in x- axis (anteroposterior) T9 (34-37 days) | -1.14 [-1.44 to -0.75]
  Left canine displacement movement in y- axis (vertical) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine displacement movement in y- axis (vertical) T9 (34-37 days) | -0.34 [-0.47 to -0.03]
  Left canine displacement movement in z- axis (transverse) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine displacement movement in z- axis (transverse) T9 (34-37 days) | -0.39 [-0.87 to -0.32]

3. Secondary Outcome: Tracking Maxillary First Molar Movement (Displacement)
Description: Magnitude of maxillary first molar tooth movement for every 4-5 days during a one month period. Measurements will be done in mm in three planes of space.
Time Frame: as for outcome 2
Population: Not all patients have data for every timepoint or side.
Measure: Median (Inter-Quartile Range); unit: Millimeters
Arm/Group | Canine retraction arm
Number analyzed (Participants) | 21
Millimeters
  Right molar displacement in x-axis (anteroposterior) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar displacement in x-axis (anteroposterior) T1 (3-5 days) | 0.03 [0.01 to 0.10]
  Right molar displacement in y-axis (vertical) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar displacement in y-axis (vertical) T1 (3-5 days) | -0.01 [-0.05 to 0.02]
  Right molar displacement in z-axis (transverse) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar displacement in z-axis (transverse) T1 (3-5 days) | -0.04 [-0.10 to 0.00]
  Left molar displacement in x-axis (anteroposterior) T1 (3-5 days): number analyzed (Participants) | 17
  Left molar displacement in x-axis (anteroposterior) T1 (3-5 days) | 0.01 [0.00 to 0.07]
  Left molar displacement in y-axis (vertical) T1 (3-5 days): number analyzed (Participants) | 17
  Left molar displacement in y-axis (vertical) T1 (3-5 days) | -0.02 [-0.04 to 0.01]
  Left molar displacement in z-axis (transverse) T1 3-5 days): number analyzed (Participants) | 17
  Left molar displacement in z-axis (transverse) T1 3-5 days) | 0.00 [-0.02 to 0.01]
  Right molar displacement movement in x- axis (anteroposterior)T2 (6-9 days): number analyzed (Participants) | 16
  Right molar displacement movement in x- axis (anteroposterior)T2 (6-9 days) | 0.03 [0.01 to 0.15]
  Right molar displacement movement in y- axis (vertical) T2 (6-9 days): number analyzed (Participants) | 16
  Right molar displacement movement in y- axis (vertical) T2 (6-9 days) | -0.09 [-0.09 to 0.00]
  Right molar displacement movement in z- axis (transverse) T2 (6-9 days): number analyzed (Participants) | 16
  Right molar displacement movement in z- axis (transverse) T2 (6-9 days) | -0.05 [-0.17 to 0.00]
  Left molar displacement movement in x- axis (anteroposterior)T2 (6-9 days): number analyzed (Participants) | 17
  Left molar displacement movement in x- axis (anteroposterior)T2 (6-9 days) | 0.02 [-0.01 to 0.11]
  Left molar displacement movement in y- axis (vertical) T2 (6-9 days): number analyzed (Participants) | 17
  Left molar displacement movement in y- axis (vertical) T2 (6-9 days) | -0.04 [-0.12 to 0.01]
  Left molar displacement movement in z- axis (transverse) T2 (6-9 days): number analyzed (Participants) | 17
  Left molar displacement movement in z- axis (transverse) T2 (6-9 days) | -0.05 [-0.17 to 0.03]
  Right molar displacement movement in x- axis (anteroposterior)T3 (10-13 days): number analyzed (Participants) | 15
  Right molar displacement movement in x- axis (anteroposterior)T3 (10-13 days) | 0.08 [0.01 to 0.17]
  Right molar displacement movement in y- axis (vertical) T3 (10-13 days): number analyzed (Participants) | 15
  Right molar displacement movement in y- axis (vertical) T3 (10-13 days) | -0.08 [-0.10 to -0.05]
  Right molar displacement movement in z- axis (transverse) T3 (10-13 days): number analyzed (Participants) | 15
  Right molar displacement movement in z- axis (transverse) T3 (10-13 days) | -0.05 [-0.12 to -0.00]
  Left molar displacement movement in x- axis (anteroposterior)T3 (10-13 days): number analyzed (Participants) | 14
  Left molar displacement movement in x- axis (anteroposterior)T3 (10-13 days) | 0.03 [-0.01 to 0.09]
  Left molar displacement movement in y- axis (vertical) T3 (10-13 days): number analyzed (Participants) | 14
  Left molar displacement movement in y- axis (vertical) T3 (10-13 days) | -0.11 [-0.13 to -0.01]
  Left molar displacement movement in z- axis (transverse) T3 (10-13 days): number analyzed (Participants) | 14
  Left molar displacement movement in z- axis (transverse) T3 (10-13 days) | -0.02 [-0.17 to 0.03]
  Right molar displacement movement in x- axis (anteroposterior)T4 (14-17 days): number analyzed (Participants) | 16
  Right molar displacement movement in x- axis (anteroposterior)T4 (14-17 days) | 0.14 [0.02 to 0.25]
  Right molar displacement movement in y- axis (vertical) T4 (14-17 days): number analyzed (Participants) | 16
  Right molar displacement movement in y- axis (vertical) T4 (14-17 days) | -0.06 [-0.14 to -0.03]
  Right molar displacement movement in z- axis (transverse) T4 (14-17 days): number analyzed (Participants) | 16
  Right molar displacement movement in z- axis (transverse) T4 (14-17 days) | -0.07 [-0.25 to -0.03]
  Left molar displacement movement in x- axis (anteroposterior)T4 (14-17 days): number analyzed (Participants) | 16
  Left molar displacement movement in x- axis (anteroposterior)T4 (14-17 days) | 0.02 [-0.06 to 0.12]
  Left molar displacement movement in y- axis (vertical) T4 (14-17 days): number analyzed (Participants) | 16
  Left molar displacement movement in y- axis (vertical) T4 (14-17 days) | -0.12 [-0.16 to -0.01]
  Left molar displacement movement in z- axis (transverse) T4 (14-17 days): number analyzed (Participants) | 16
  Left molar displacement movement in z- axis (transverse) T4 (14-17 days) | -0.14 [-0.20 to 0.06]
  Right molar displacement movement in x- axis (anteroposterior)T5 (18-21 days): number analyzed (Participants) | 15
  Right molar displacement movement in x- axis (anteroposterior)T5 (18-21 days) | 0.15 [0.00 to 0.25]
  Right molar displacement movement in y- axis (vertical) T5 (18 -21days): number analyzed (Participants) | 15
  Right molar displacement movement in y- axis (vertical) T5 (18 -21days) | -0.10 [-0.18 to 0.0]
  Right molar displacement movement in z- axis (transverse) T5 (18-21 days): number analyzed (Participants) | 15
  Right molar displacement movement in z- axis (transverse) T5 (18-21 days) | -0.09 [-0.26 to -0.02]
  Left molar displacement movement in x- axis (anteroposterior)T5 (18-21 days): number analyzed (Participants) | 15
  Left molar displacement movement in x- axis (anteroposterior)T5 (18-21 days) | 0.04 [-0.04 to 0.18]
  Left molar displacement movement in y- axis (vertical) T5 (18-21 days): number analyzed (Participants) | 15
  Left molar displacement movement in y- axis (vertical) T5 (18-21 days) | -0.12 [-0.16 to -0.06]
  Left molar displacement movement in z- axis (transverse) T5 (18-21 days): number analyzed (Participants) | 15
  Left molar displacement movement in z- axis (transverse) T5 (18-21 days) | -0.09 [-0.23 to 0.07]
  Right molar displacement movement in x- axis (anteroposterior)T6 (22-25 days): number analyzed (Participants) | 13
  Right molar displacement movement in x- axis (anteroposterior)T6 (22-25 days) | 0.13 [0.07 to 0.24]
  Right molar displacement movement in y- axis (vertical) T6 (22-25 days): number analyzed (Participants) | 13
  Right molar displacement movement in y- axis (vertical) T6 (22-25 days) | -0.09 [-0.18 to 0.03]
  Right molar displacement movement in z- axis (transverse) T6 (22 -25 days): number analyzed (Participants) | 13
  Right molar displacement movement in z- axis (transverse) T6 (22 -25 days) | -0.13 [-0.32 to -0.06]
  Left molar displacement movement in x- axis (anteroposterior)T6 (22-25 days): number analyzed (Participants) | 15
  Left molar displacement movement in x- axis (anteroposterior)T6 (22-25 days) | -0.02 [-0.09 to 0.09]
  Left molar displacement movement in y- axis (vertical) T6 (22-25 days): number analyzed (Participants) | 15
  Left molar displacement movement in y- axis (vertical) T6 (22-25 days) | -0.15 [-0.20 to -0.05]
  Left molar displacement movement in z- axis (transverse) T6 (22-25 days): number analyzed (Participants) | 15
  Left molar displacement movement in z- axis (transverse) T6 (22-25 days) | -0.04 [-0.32 to 0.13]
  Right molar displacement movement in x- axis (anteroposterior)T7 (26-29 days): number analyzed (Participants) | 17
  Right molar displacement movement in x- axis (anteroposterior)T7 (26-29 days) | 0.25 [0.11 to 0.41]
  Right molar displacement movement in y- axis (vertical) T7 (26-29 days): number analyzed (Participants) | 17
  Right molar displacement movement in y- axis (vertical) T7 (26-29 days) | -0.14 [-0.21 to 0.04]
  Right molar displacement movement in z- axis (transverse) T7 (26-29 days): number analyzed (Participants) | 17
  Right molar displacement movement in z- axis (transverse) T7 (26-29 days) | -0.05 [-0.27 to 0.01]
  Left molar displacement movement in x- axis (anteroposterior)T7 (26-29 days): number analyzed (Participants) | 17
  Left molar displacement movement in x- axis (anteroposterior)T7 (26-29 days) | 0.08 [-0.05 to 0.18]
  Left molar displacement movement in y- axis (vertical) T7 (26-29 days): number analyzed (Participants) | 17
  Left molar displacement movement in y- axis (vertical) T7 (26-29 days) | -0.16 [-0.25 to -0.03]
  Left molar displacement movement in z- axis (transverse) T7 (26-29 days): number analyzed (Participants) | 17
  Left molar displacement movement in z- axis (transverse) T7 (26-29 days) | -0.11 [-0.28 to 0.08]
  Right molar displacement movement in x- axis (anteroposterior)T8 (30-33 days): number analyzed (Participants) | 10
  Right molar displacement movement in x- axis (anteroposterior)T8 (30-33 days) | 0.23 [0.08 to 0.34]
  Right molar displacement movement in y- axis (vertical) T8 (30-33 days): number analyzed (Participants) | 10
  Right molar displacement movement in y- axis (vertical) T8 (30-33 days) | -0.10 [-0.20 to -0.01]
  Right molar displacement movement in z- axis (transverse) T8 (30-33 days): number analyzed (Participants) | 10
  Right molar displacement movement in z- axis (transverse) T8 (30-33 days) | -0.19 [-0.33 to -0.10]
  Left molar displacement movement in x- axis (anteroposterior)T8 (30-33 days): number analyzed (Participants) | 11
  Left molar displacement movement in x- axis (anteroposterior)T8 (30-33 days) | 0.00 [-0.14 to 0.12]
  Left molar displacement movement in y- axis (vertical) T8 (30-33 days): number analyzed (Participants) | 11
  Left molar displacement movement in y- axis (vertical) T8 (30-33 days) | -0.19 [-0.32 to -0.16]
  Left molar displacement movement in z- axis (transverse) T8 (30-33 days): number analyzed (Participants) | 11
  Left molar displacement movement in z- axis (transverse) T8 (30-33 days) | -0.13 [-0.38 to 0.05]
  Right molar displacement movement in x- axis (anteroposterior)T9 (34-37 days): number analyzed (Participants) | 7
  Right molar displacement movement in x- axis (anteroposterior)T9 (34-37 days) | 0.34 [0.20 to 0.41]
  Right molar displacement movement in y- axis (vertical) T9 (34-37 days): number analyzed (Participants) | 7
  Right molar displacement movement in y- axis (vertical) T9 (34-37 days) | -0.07 [-0.19 to -0.06]
  Right molar displacement movement in z- axis (transverse) T9 (34-37 days): number analyzed (Participants) | 7
  Right molar displacement movement in z- axis (transverse) T9 (34-37 days) | -0.17 [-0.36 to -0.03]
  Left molar displacement movement in x- axis (anteroposterior)T9 (34-37 days): number analyzed (Participants) | 9
  Left molar displacement movement in x- axis (anteroposterior)T9 (34-37 days) | -0.01 [-0.05 to 0.10]
  Left molar displacement movement in y- axis (vertical) T9 (34-37 days): number analyzed (Participants) | 9
  Left molar displacement movement in y- axis (vertical) T9 (34-37 days) | -0.15 [-0.23 to -0.10]
  Left molar displacement movement in z- axis (transverse) T9 (34 -37 days): number analyzed (Participants) | 9
  Left molar displacement movement in z- axis (transverse) T9 (34 -37 days) | -0.02 [-0.20 to 0.17]

4. Secondary Outcome: Tracking Maxillary Canine Tooth Movement (Rotation)
Description: Magnitude of canine tooth movement for every 4-5 days during a one month period. Measurements will be done in degrees in three planes of space.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Canine retraction arm
Number analyzed (Participants) | 21
degrees
  Right canine rotational movement (x -axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right canine rotational movement (x -axis) T1 (3-5 days) | 0.19 [-0.13 to 0.52]
  Right canine rotational movement (y -axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right canine rotational movement (y -axis) T1 (3-5 days) | -0.34 [-0.83 to 0.13]
  Right canine rotational movement (z-axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right canine rotational movement (z-axis) T1 (3-5 days) | 0.02 [-0.35 to 0.27]
  Left canine rotational movement (x -axis) T1 (3-5 days): number analyzed (Participants) | 17
  Left canine rotational movement (x -axis) T1 (3-5 days) | -0.01 [-0.25 to 0.15]
  Left canine rotational movement (y -axis) T1 (3-5 days): number analyzed (Participants) | 17
  Left canine rotational movement (y -axis) T1 (3-5 days) | -0.66 [-3.45 to -0.05]
  Left canine rotational movement (z -axis) T1 3-5 days): number analyzed (Participants) | 17
  Left canine rotational movement (z -axis) T1 3-5 days) | 0.06 [-0.17 to 0.21]
  Right canine rotational movement (x -axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right canine rotational movement (x -axis) T2 (6-9 days) | 0.00 [-0.28 to 0.57]
  Right canine rotational movement (y -axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right canine rotational movement (y -axis) T2 (6-9 days) | -1.64 [-2.9 to -0.88]
  Right canine rotational movement (z-axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right canine rotational movement (z-axis) T2 (6-9 days) | -0.07 [-0.68 to 0.32]
  Left canine rotational movement (x -axis) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine rotational movement (x -axis) T2 (6-9 days) | -0.20 [-0.36 to 0.05]
  Left canine rotational movement (y -axis) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine rotational movement (y -axis) T2 (6-9 days) | -2.28 [-3.50 to -0.55]
  Left canine rotational movement (z -axis) T2 (6-9 days): number analyzed (Participants) | 17
  Left canine rotational movement (z -axis) T2 (6-9 days) | -0.36 [-0.78 to 0.00]
  Right canine rotational movement (x -axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right canine rotational movement (x -axis) T3 (10-13 days) | 0.04 [-0.10 to 0.31]
  Right canine rotational movement (y -axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right canine rotational movement (y -axis) T3 (10-13 days) | -2.14 [-4.39 to -0.69]
  Right canine rotational movement (z-axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right canine rotational movement (z-axis) T3 (10-13 days) | -0.28 [-1.14 to 0.61]
  Left canine rotational movement (x -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine rotational movement (x -axis) T3 (10-13 days) | -0.32 [-1.01 to 0.09]
  Left canine rotational movement (y -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine rotational movement (y -axis) T3 (10-13 days) | -1.23 [-3.34 to 0.06]
  Left canine rotational movement (z -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left canine rotational movement (z -axis) T3 (10-13 days) | -0.82 [-1.12 to -0.23]
  Right canine rotational movement (x -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right canine rotational movement (x -axis) T4 (14-17 days) | -0.24 [-0.76 to 0.05]
  Right canine rotational movement (y -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right canine rotational movement (y -axis) T4 (14-17 days) | -2.23 [-4.29 to -1.15]
  Right canine rotational movement (z-axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right canine rotational movement (z-axis) T4 (14-17 days) | -0.47 [-1.69 to -0.10]
  Left canine rotational movement (x -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine rotational movement (x -axis) T4 (14-17 days) | -0.38 [-1.04 to -0.24]
  Left canine rotational movement (y -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine rotational movement (y -axis) T4 (14-17 days) | -2.19 [-4.38 to -0.64]
  Left canine rotational movement (z -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left canine rotational movement (z -axis) T4 (14-17 days) | -0.91 [-1.40 to -0.56]
  Right canine rotational movement (x -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right canine rotational movement (x -axis) T5 (18-21 days) | -0.52 [-1.25 to -0.02]
  Right canine rotational movement (y-axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right canine rotational movement (y-axis) T5 (18-21 days) | -3.06 [-4.56 to -1.95]
  Right canine rotational movement (z -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right canine rotational movement (z -axis) T5 (18-21 days) | -0.82 [-1.48 to -0.28]
  Left canine rotational movement (x -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left canine rotational movement (x -axis) T5 (18-21 days) | -0.69 [-1.44 to -0.16]
  Left canine rotational movement (y -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left canine rotational movement (y -axis) T5 (18-21 days) | -3.75 [-3.97 to -0.78]
  Left canine rotational movement (z -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left canine rotational movement (z -axis) T5 (18-21 days) | -0.97 [-1.99 to -0.39]
  Right canine rotational movement (x -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right canine rotational movement (x -axis) T6 (22-25 days) | -0.72 [-1.02 to -0.15]
  Right canine rotational movement (y -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right canine rotational movement (y -axis) T6 (22-25 days) | -3.61 [-6.09 to -2.14]
  Right canine rotational movement (z -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right canine rotational movement (z -axis) T6 (22-25 days) | -1.51 [-1.82 to -0.74]
  Left canine rotational movement (x -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine rotational movement (x -axis) T6 (22-25 days) | -0.80 [-1.19 to -0.15]
  Left canine rotational movement (y -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine rotational movement (y -axis) T6 (22-25 days) | -3.76 [-6.39 to -1.34]
  Left canine rotational movement (z -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left canine rotational movement (z -axis) T6 (22-25 days) | -1.04 [-2.00 to -0.53]
  Right canine rotational movement (x -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine rotational movement (x -axis) T7 (26-29 days) | -0.41 [-1.59 to -0.08]
  Right canine rotational movement (y -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine rotational movement (y -axis) T7 (26-29 days) | -3.50 [-4.63 to -1.94]
  Right canine rotational movement (z -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Right canine rotational movement (z -axis) T7 (26-29 days) | -1.18 [-1.65 to -0.33]
  Left canine rotational movement (x -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine rotational movement (x -axis) T7 (26-29 days) | -0.76 [-1.24 to -0.13]
  Left canine rotational movement (y-axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine rotational movement (y-axis) T7 (26-29 days) | -2.93 [-6.47 to -1.54]
  Left canine rotational movement (z -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left canine rotational movement (z -axis) T7 (26-29 days) | -1.29 [-1.87 to -0.71]
  Right canine rotational movement (x -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine rotational movement (x -axis) T8 (30-33 days) | -1.04 [-2.01 to -0.18]
  Right canine rotational movement (y -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine rotational movement (y -axis) T8 (30-33 days) | -3.67 [-4.53 to -2.10]
  Right canine rotational movement (z -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right canine rotational movement (z -axis) T8 (30-33 days) | -1.16 [-1.41 to 0.04]
  Left canine rotational movement (x -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine rotational movement (x -axis) T8 (30-33 days) | -0.77 [-1.43 to -0.13]
  Left canine rotational movement (y -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine rotational movement (y -axis) T8 (30-33 days) | -4.17 [-7.86 to -2.47]
  Left canine rotational movement (z -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left canine rotational movement (z -axis) T8 (30-33 days) | -2.23 [-2.68 to -0.42]
  Right canine rotational movement (x -axis) T9 (34-37 days): number analyzed (Participants) | 7
  Right canine rotational movement (x -axis) T9 (34-37 days) | -0.43 [-1.74 to 0.35]
  Right canine rotational movement (y -axis) T9 (34-7 days): number analyzed (Participants) | 7
  Right canine rotational movement (y -axis) T9 (34-7 days) | -3.96 [-5.03 to -2.96]
  Right canine rotational movement (z -axis) T9 (34-37 days): number analyzed (Participants) | 7
  Right canine rotational movement (z -axis) T9 (34-37 days) | -1.67 [-2.02 to -0.60]
  Left canine rotational movement (x -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine rotational movement (x -axis) T9 (34-37 days) | -0.72 [-1.46 to -0.26]
  Left canine rotational movement (y -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine rotational movement (y -axis) T9 (34-37 days) | -3.06 [-7.05 to -3.00]
  Left canine rotational movement (z -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left canine rotational movement (z -axis) T9 (34-37 days) | -0.71 [-1.61 to -0.12]

5. Secondary Outcome: Tracking Maxillary First Molar Displacement (Rotation)
Description: Magnitude of maxillary first molar tooth movement for every 4-5 days during a one month period. Measurements will be done in degrees in three planes of space.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Canine retraction arm
Number analyzed (Participants) | 21
Degrees
  Right molar rotational movement (x-axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar rotational movement (x-axis) T1 (3-5 days) | -0.06 [-0.36 to 0.05]
  Right molar rotational movement (y-axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar rotational movement (y-axis) T1 (3-5 days) | 0.00 [-0.28 to 0.30]
  Right molar rotational movement (z-axis) T1 (3-5 days): number analyzed (Participants) | 17
  Right molar rotational movement (z-axis) T1 (3-5 days) | -0.00 [-0.24 to 0.28]
  Left molar rotational movement (x-axis) T1 3-5 days): number analyzed (Participants) | 17
  Left molar rotational movement (x-axis) T1 3-5 days) | 0.02 [-0.18 to 0.23]
  Left molar rotational movement (y-axis)T1 (3-5 days): number analyzed (Participants) | 17
  Left molar rotational movement (y-axis)T1 (3-5 days) | 0.20 [0.00 to 0.39]
  Left molar rotational movement (z-axis) T1 (3-5 days): number analyzed (Participants) | 17
  Left molar rotational movement (z-axis) T1 (3-5 days) | 0.00 [-0.18 to 0.11]
  Right molar rotational movement (x -axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right molar rotational movement (x -axis) T2 (6-9 days) | -0.14 [-0.40 to 0.01]
  Right molar rotational movement (y -axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right molar rotational movement (y -axis) T2 (6-9 days) | 0.05 [-0.22 to 0.54]
  Right molar rotational movement (z -axis) T2 (6-9 days): number analyzed (Participants) | 16
  Right molar rotational movement (z -axis) T2 (6-9 days) | 0.00 [-0.44 to 0.82]
  Left molar rotational movement (x -axis) T2 (6-9 days): number analyzed (Participants) | 18
  Left molar rotational movement (x -axis) T2 (6-9 days) | 0.03 [-0.03 to 0.23]
  Left molar rotational movement (y -axis) T2 (6-9 days): number analyzed (Participants) | 18
  Left molar rotational movement (y -axis) T2 (6-9 days) | 0.55 [0.15 to 0.97]
  Left molar rotational movement (z -axis) T2 (6-9 days): number analyzed (Participants) | 18
  Left molar rotational movement (z -axis) T2 (6-9 days) | 0.11 [-0.31 to 0.42]
  Right molar rotational movement (x -axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right molar rotational movement (x -axis) T3 (10-13 days) | -0.46 [-0.85 to 0.08]
  Right molar rotational movement (y -axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right molar rotational movement (y -axis) T3 (10-13 days) | 0.24 [-0.28 to 0.69]
  Right molar rotational movement (z -axis) T3 (10-13 days): number analyzed (Participants) | 15
  Right molar rotational movement (z -axis) T3 (10-13 days) | -0.07 [-0.55 to 0.37]
  Left molar rotational movement (x -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left molar rotational movement (x -axis) T3 (10-13 days) | 0.20 [-0.16 to 0.39]
  Left molar rotational movement (y -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left molar rotational movement (y -axis) T3 (10-13 days) | 0.44 [0.20 to 0.87]
  Left molar rotational movement (z -axis) T3 (10-13 days): number analyzed (Participants) | 14
  Left molar rotational movement (z -axis) T3 (10-13 days) | 0.24 [-0.22 to 1.17]
  Right molar rotational movement (x -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right molar rotational movement (x -axis) T4 (14-17 days) | -0.48 [-0.76 to -0.31]
  Right molar rotational movement (y -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right molar rotational movement (y -axis) T4 (14-17 days) | 0.52 [-0.27 to 1.70]
  Right molar rotational movement (z -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Right molar rotational movement (z -axis) T4 (14-17 days) | 0.21 [-0.26 to 0.54]
  Left molar rotational movement (x -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left molar rotational movement (x -axis) T4 (14-17 days) | -0.24 [-0.40 to 0.38]
  Left molar rotational movement (y -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left molar rotational movement (y -axis) T4 (14-17 days) | 0.62 [0.30 to 1.02]
  Left molar rotational movement (z -axis) T4 (14-17 days): number analyzed (Participants) | 16
  Left molar rotational movement (z -axis) T4 (14-17 days) | 0.11 [-0.42 to 0.63]
  Right molar rotational movement (x -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right molar rotational movement (x -axis) T5 (18-21 days) | -0.13 [-0.58 to 0.36]
  Right molar rotational movement (y -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right molar rotational movement (y -axis) T5 (18-21 days) | 1.46 [0.07 to 2.13]
  Right molar rotational movement (z -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Right molar rotational movement (z -axis) T5 (18-21 days) | 0.53 [-0.20 to 0.91]
  Left molar rotational movement (x -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left molar rotational movement (x -axis) T5 (18-21 days) | -0.11 [-0.42 to 0.75]
  Left molar rotational movement (y -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left molar rotational movement (y -axis) T5 (18-21 days) | 0.94 [0.78 to 2.35]
  Left molar rotational movement (z -axis) T5 (18-21 days): number analyzed (Participants) | 15
  Left molar rotational movement (z -axis) T5 (18-21 days) | 0.26 [-0.65 to 0.86]
  Right molar rotational movement (x -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right molar rotational movement (x -axis) T6 (22-25 days) | -0.34 [-0.82 to 0.65]
  Right molar rotational movement (y -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right molar rotational movement (y -axis) T6 (22-25 days) | 0.59 [-0.75 to 2.95]
  Right molar rotational movement (z -axis) T6 (22-25 days): number analyzed (Participants) | 13
  Right molar rotational movement (z -axis) T6 (22-25 days) | 0.07 [-0.35 to 0.83]
  Left molar rotational movement (x -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left molar rotational movement (x -axis) T6 (22-25 days) | 0.49 [-0.36 to 0.96]
  Left molar rotational movement (y -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left molar rotational movement (y -axis) T6 (22-25 days) | 1.46 [0.81 to 2.11]
  Left molar rotational movement (z -axis) T6 (22-25 days): number analyzed (Participants) | 15
  Left molar rotational movement (z -axis) T6 (22-25 days) | 0.76 [-0.24 to 1.23]
  Righ molar rotational movement (x -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Righ molar rotational movement (x -axis) T7 (26-29 days) | -0.35 [-0.89 to 0.23]
  Right molar rotational movement (y -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Right molar rotational movement (y -axis) T7 (26-29 days) | 1.31 [-0.68 to 3.06]
  Right molar rotational movement (z -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Right molar rotational movement (z -axis) T7 (26-29 days) | 0.39 [0.00 to 1.28]
  Left molar rotational movement (x -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left molar rotational movement (x -axis) T7 (26-29 days) | 0.20 [-0.38 to 0.99]
  Left molar rotational movement (y -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left molar rotational movement (y -axis) T7 (26-29 days) | 1.53 [1.13 to 2.56]
  Left molar rotational movement (z -axis) T7 (26-29 days): number analyzed (Participants) | 17
  Left molar rotational movement (z -axis) T7 (26-29 days) | 0.41 [-1.01 to 1.25]
  Right molar rotational movement (x -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right molar rotational movement (x -axis) T8 (30-33 days) | -0.59 [-0.97 to -0.14]
  Right molar rotational movement (y -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right molar rotational movement (y -axis) T8 (30-33 days) | 1.93 [0.31 to 3.24]
  Right molar rotational movement (z -axis) T8 (30-33 days): number analyzed (Participants) | 10
  Right molar rotational movement (z -axis) T8 (30-33 days) | 0.98 [0.16 to 1.45]
  Left molar rotational movement (x -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left molar rotational movement (x -axis) T8 (30-33 days) | -0.01 [-0.93 to 0.33]
  Left molar rotational movement (y -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left molar rotational movement (y -axis) T8 (30-33 days) | 1.78 [0.36 to 3.33]
  Left molar rotational movement (z -axis) T8 (30-33 days): number analyzed (Participants) | 11
  Left molar rotational movement (z -axis) T8 (30-33 days) | 0.45 [-0.05 to 1.22]
  Right molar rotational movement (x -axis) T9 (34-37 days): number analyzed (Participants) | 7
  Right molar rotational movement (x -axis) T9 (34-37 days) | 3.13 [-0.04 to 3.29]
  Right molar rotational movement (y-axis) T9 (34-37 days): number analyzed (Participants) | 7
  Right molar rotational movement (y-axis) T9 (34-37 days) | 0.57 [0.13 to 1.08]
  Right molar rotational movement (z -axis) T9 (34-37 days): number analyzed (Participants) | 7
  Right molar rotational movement (z -axis) T9 (34-37 days) | 0.77 [0.07 to 1.34]
  Left molar rotational movement (x -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left molar rotational movement (x -axis) T9 (34-37 days) | 0.60 [-0.64 to 0.68]
  Left molar rotational movement (y -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left molar rotational movement (y -axis) T9 (34-37 days) | 2.67 [1.29 to 4.35]
  Left molar rotational movement (z -axis) T9 (34-37 days): number analyzed (Participants) | 9
  Left molar rotational movement (z -axis) T9 (34-37 days) | 0.97 [0.42 to 1.07]

ADVERSE EVENTS:
Time Frame: For each subject up to 1 month of their participation in the study.
Description: Adverse Event Reporting was conducted in accordance with the Institutional Review Board (IRB) protocol at the University of Connecticut Health Center (21-113-2). Adverse event data collected systematically per set times in subject recruitment. During the study, there were a total of 6 meetings.
Arm/Group | Canine retraction arm
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05780788/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05780788/ICF_001.pdf